CLINICAL TRIAL: NCT06256172
Title: Medlink for Diagnosing of Diabetes Mellitus, COPD, CHF, Myasthenia Gravis and Hypertension
Acronym: Medlink
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olawuyi Racett Nigeria Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: M101
Record Dates: First submitted 2024-01-11; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus; Chronic Obstructive Pulmonary Disease; Congestive Heart Failure; Myasthenia Gravis; Hypertension
MeSH Terms: conditions — Diabetes Mellitus; Pulmonary Disease, Chronic Obstructive; Heart Failure; Myasthenia Gravis; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medlink RPM (Experimental): The 10 Patients enrolled in this arm tested the ue of Medlink in Measuring and reporting their Physiological Paramters in Oder to remotely obtain access to health care for the following diseases: Myasthenia Gravis, Hypertension, Chronic Heart Failure, Diabetes Mellitus, and Chronic Obstruction Pulmonary Disorder.
  Interventions: Device: Medlink

INTERVENTIONS:
Device: Medlink — The 10 Patients enrolled in this arm tested the ue of Medlink in Measuring and reporting their Physiological Paramters in Oder to remotely obtain access to health care for the following diseases: Myasthenia Gravis, Hypertension, Chronic Heart Failure, Diabetes Mellitus, and Chronic Obstruction Pulmonary Disorder.

SUMMARY:
MEDLINK IS A POCKET-SIZED MEDLINK is a pocket-sized, verbally interactive, programmable medical device that allows physicians to select which medical measurements they would like to take for a specific patient. The Physiological Parameters that can be measured by MEDLINK include, but is not limited to: Electrocardiography (ECG), Blood Pressure, Heart Rate, Blood Glucose, Pulse Rate, Blood Oxygen Saturation (SPO2), Electromyography (EMG) body temperature, and Respiratory Data. MEDLINK is a pocket-sized, verbally interactive, programmable medical device that allows physicians to select which medical measurements they would like to take for a specific patient.

When the patient takes MEDLINK home and switches it on, the device verbally guides the patient to acquire the measurements requested by the his or her physician.

This information is transmitted to the physican's email for medical analysis, check up and/or follow up.

This Study was executed by TWO (2) MEDICAL CONSULTANTS: Dr. Michael Olawuyi (mgolawuyi@gmail.com) and Dr, Matthew Olawuyi (olawuyiracettnigerialtd@outlook.com)

DETAILED DESCRIPTION:
MEDLINK is a pocket-sized, verbally interactive, programmable medical device that allows physicians to select which medical measurements they would like to take for a specific patient. The Physiological Parameters that can be measured by MEDLINK include, but is not limited to: Electrocardiography (ECG), Blood Pressure, Heart Rate, Blood Glucose, Pulse Rate, Blood Oxygen Saturation (SPO2), Electromyography (EMG) body temperature, and Respiratory Data. After programming of the device by the Physician, MEDLINK can be given to the desired patient to take home for Remote Patient Monitoring (RPM).

When the patient switches on the device at home, MEDLINK verbally guides the patient to acquire the measurements requested by his or her Physician. This information is automatically and wirelessly transmitted to the Physician's Mobile Phone and Email Address for medical analysis, check up, and/or follow up. MEDLINK has its own software application that allows the Physician to view and analyse the measured Physiological Parameters for any Patient. MEDLINK also has the potential to allow Patient-Physician Communication during the RPM Period.

One of the key innovations of MEDLINK is that it is able to acquire a diverse range of physiological parameters. This makes it useful to physicians in different areas of specialization in the medical field. In addition to this, MEDLINK also accurately measures all Physiological Parameters of the Patient through a single digit finger being inserted into the appropriate position in the pocket-device, making it extremely easy to use. MEDLINK is the first medical device that performs blood glucose measurement using Infrared Technology, as opposed to the standardized lancet finger-pricking technology.

MEDLINK allows Physicians in any specialization to monitor patients outside of the hospital setting for as long as is needed. It can be used to monitor patients after they have been discharged from the hospital. It also allows individuals to have quality access to basic health care.

Ten Patients were recruited for this Study and tested the use of MEDLINK in measuring physiological parameters and providing remote access to basic health care.

This Study was executed by TWO (2) MEDICAL CONSULTANTS: Dr. Michael Olawuyi (mgolawuyi@gmail.com) and Dr, Matthew Olawuyi (olawuyiracettnigerialtd@outlook.com)

ELIGIBILITY:
Inclusion Criteria:

* NONE

Exclusion Criteria:

* NONE

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2023-12-16 (Actual); Study Completion 2023-12-16 (Actual)

PRIMARY OUTCOMES:
Electrocardiography (ECG) (1 PQRS Interval acquired) using the ECG unit in Medlink | Measurement is done Once daily for 2 weeks
  1 PQRS Interval is acquired.
5 readings of Blood Pressure (Systolic and Diastolic Pressure) in mmHg using the Blood Pressure unit in Medlink is acquired and the average value is reported | Measurement is done Once daily for 2 weeks
  Acquisition of 5 readings of Blood Pressure (Systolic and Diastolic Pressure) in mmHg and the average value is reported
5 readings of 1 beat of Heart Rate in bpm is acquired using the Heart Rate unit in Medlink and the average value is reported. | Measurement is done Once daily for 2 weeks
  Acquisition of 5 readings of Heart Rate in bpm and the average vallue is reported
5 readings of Blood Glucose in mmol/L using the Infrared Glucometer unit in Medlink is acquired and the average value is reported | Measurement is done Once daily for 2 weeks
  Acquisition of 5 readings of Blood Glucose in mmol/L and the average value is reported
5 readings of Pulse in bpm using the Pulse Rate unit in Medlink and the average value is reported | Measurement is done Once daily for 2 weeks
  Acquisition of 5 readings of Pulse in bpm and the average value is reported
5 readings of SPO2 in percent using the SPO2 unit in Medlink and the average value is reported | Measurement is done Once daily for 2 weeks
  Acquisition of 5 readings of SPO2 or Blood Oxygen Saturation and the average value is reported
5 readings of Electromyography (EMG) Power in Analog Values in the Beta Band is measured using the EMG unit in Medlink and the average value is reported | Measurement is done Once daily for 2 weeks
  Acquisition of 5 readings of Electromyography or Muscle Strength Power in the Beta band and the average value is reported
5 readings of Body Temperature in Degrees Celcius using the Body Temperature Unit of Medlink and the average value is reported. | Measurement is done Once daily for 2 weeks
  Acquisition of 5 readings of Body Temperature in Degrees Celcius and the average value is reported
5 readings of Respiratory Data (FEV1, FVC, FEV1/FVC ratio) in L using the Respiratory unit in Medlink is acquired and the average value is reported. | Measurement is done Once daily for 2 weeks
  Acquisition of 5 readings of Respiratory Data (FEV1, FVC, FEV1/FVC ratio) in L and the average value is reported

CONTACTS AND LOCATIONS:
Overall Officials: Michael Olawuyi, MPH, Study Director — Olawuyi Racett Nigeria Ltd. United Kingdom RC14668218; Matthew Olawuyi, MBBS, Study Chair — Olawuyi Racett Nigeria Ltd. United Kingdom RC14668218; Esther Olawuyi, D.Sc., Principal Investigator — Olawuyi Racett Nigeria Ltd. United Kingdom RC14668218
Locations (1):
- Olawuyi Racett Nigeria Ltd., London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data Gathered from the Trial will be made available through Certified Publications
Supporting Information: CSR
Time Frame: Data is available as of 20/01/2024 until 20/01/2034
Access Criteria: Data is available to all the public

DOCUMENTS (1):
  • Study Protocol (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT06256172/Prot_000.pdf